CLINICAL TRIAL: NCT04622436
Title: Comparison of MicroStream Capnography and Pulseoxymeter in Sedation of Pediatric Patients Undergoing Magnetic Resonance Imaging
Brief Title: Early Recognition of Hypoxia in Pediatric Patient Sedation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Canan Yılmaz, Department of Anesthesiology and Reanimation Director, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-25 2020/09-03
Record Dates: First submitted 2020-10-16; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Desaturation of Blood
Keywords: Hypoxia; Desaturation; MicroStream Capnography; Pulseoxymeter
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early recognition of hypoxia through monitoring in sedation practices in pediatric patients

DETAILED DESCRIPTION:
In pediatric Magnetic Resonance Imaging, sedation is applied to pediatric patients of all age groups from newborn to adolescence in order to prevent the anxiety and movement of the patients during the imaging. It was aimed to compare the capnograph and pulse oximeter used for early detection of hypoxia in patient follow-up and to monitor the depth of sedation with the sedation score in the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 18 years of age who underwent magnetic resonance imaging with sedoanalgesia

Exclusion Criteria:

* Patients over the age of 18,
* Those who do not speak Turkish,
* Presence of deformities in the nose and forehead,
* Those with nail polish and henna on their nails

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients under ages 18
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Early recognition of hypoxia | during the procedure
  The rapid recognition of hypoxia that may occur with the initiation of the procedure
the changes in partial oxygen saturation | during the procedure
  The rapid recognition of changes in partial oxygen saturation

SECONDARY OUTCOMES:
Sedation score | during the procedure
  Monitoring ramsey sedation scale. The minimum value is 1 and the maximum value is 6. Higher score means more sedatized.
recovery time | immediately after the procedure
  length of stay in the recovery room

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yuksek Ihtisas Education and Research Hospital, Bursa, Yıldırım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided